CLINICAL TRIAL: NCT01564810
Title: Study of Cetuximab in Combination With Chemotherapy for the First Treatment of Metastatic Colorectal Cancer
Brief Title: Cetuximab in Combination With Chemotherapy for the Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Jianmin Xu, PhD Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-03
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms
Keywords: liver metastasis; colorectal cancer; cetuximab; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): patients received cetuximab in combination with chemotherapy
  Interventions: Drug: Cetuximab; Drug: chemotherapy of mFOLFOX6 or FOLFIRI
- Arm B (Active Comparator): Patients received chemotherapy (mFOLFOX6 or FOLFIRI) alone. mFOLFOX6 (day 1, oxaliplatin 85 mg/m², folinic acid 400 mg/m², and fluorouracil 400 mg/m² intravenous bolus, then 2400 mg/m² over 46 h continuous infusion) FOLFIRI (day 1, irinotecan 180mg/m2, folinic acid 400 mg/m², and fluorouracil 400 mg/m² intravenous bolus, then continuous infusion for 46 hours of 2400 mg/m2).
  Interventions: Drug: chemotherapy of mFOLFOX6 or FOLFIRI

INTERVENTIONS:
Drug: Cetuximab — On day 1 of a 14 day treatment cycle, patients received a 2-hour infusion of cetuximab (initial dose 400 mg/m2 in week 1, and 250 mg/m2 weekly during 1 hour thereafter) followed after 1 hour by chemotherapy of FOLFOX or FOLFIRI until progressive disease or unacceptable toxicity.
  Other Names: Erbitux
  Arms: Arm A
Drug: chemotherapy of mFOLFOX6 or FOLFIRI — FOLFOX-4 (oxaliplatin, 85mg/m2 on day 1 infused during 2 hours;LV200mg/m2ondays 1and 2 infused during 2 hours, together with or following oxaliplatin; followed by FU 400 mg/m2 intravenous bolus then 600 mg/m2 intravenous infusion over 22 hours on days 1 and 2) FOLFIRI(irinotecan 180mg/m2 on day 1 infused during 2 hours; fluorouracil in a bolus of 400 mg/m2 and then continuous infusion for 46 hours of 2400 mg/m2)
  Other Names: mFOLFOX6

SUMMARY:
In this study, the investigators assessed the effect of Cetuximab in combination with chemotherapy in the treatment of unresectable metastatic colorectal cancer.

DETAILED DESCRIPTION:
Patients will be eligible for inclusion if their primary tumors have been resected and if the patients have histologically confirmed wild-type-KRAS colorectal adenocarcinoma with synchronous liver-confined metastases deemed non-resectable. Eligible patients will be randomly assigned to chemotherapy plus cetuximab (arm A) or chemotherapy alone (arm B). Treatment will be planned to commence between 2 and 4 weeks after the primary surgery. Treatment will continue until tumor response indicates suitability for surgery for liver metastases or until disease progression or unacceptable toxic effects. The primary endpoint is the conversion rate to radical resection for liver metastases，which will be assessed by local multidisciplinary team (includes more than three liver surgeons and one radiologist) with the use of contrast-enhanced CT or MRI after 4 cycles and then every other 2 cycles up to 12 cycles. To provide an objective assessment of changes in resectability, radiological images will be presented by a radiologist to more than 3 liver surgeons, who are blinded to the clinical data. Patients will be considered resectable if 50% or more of surgeons vote for radical resection of LM. For patients whose liver-metastases are assessed resectable, resection should be scheduled to be performed within 2~3 weeks of the last treatment cycle. Following resection, patients will be advised to continue the same therapeutic regimen until the treatments reach a sum of 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumour has undergone radical resection and histologically confirmed colorectal adenocarcinoma;
3. Together with clinical or radiological evidence of first occurrence of non-resectable synchronous liver-only metastases
4. With evidence of tumor EGFR expression and KRAS gene wild-type status;
5. With one measurable tumor.
6. Performance status (ECOG) 0~1
7. A life expectancy of ≥ 3 months
8. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization)
9. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either AST or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
10. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Previous exposure to target therapy, chemotherapy, radiotherapy or intervention therapy for colorectal liver metastases.
2. Known or suspected extrahepatic metastases.
3. Patients with known hypersensitivity reactions to any of the components of the study treatments.
4. Having previously participated in a study which included a possibility of being allocated to cetuximab therapy (whether or not the patient actually received cetuximab)
5. Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or left ventricular ejection fraction (LVEF) below the institutional range of normal
6. Acute or sub-acute intestinal occlusion
7. Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
8. Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
9. Known drug abuse/ alcohol abuse
10. Legal incapacity or limited legal capacity
11. Pre-existing peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-09; Primary Completion 2012-06 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
the rate of patients converted to resection for liver metastases | 3 years
  To explore whether cetuximab in combination with chemotherapy as treatment could improve the resection rate in patients with KRAS wild-type, unresectable colorectal liver-limited metastases compared with chemotherapy alone.

SECONDARY OUTCOMES:
progression free survival | 3 years
  PFS will be defined as the period from the first day of cetuximab treatment or chemotherapy to the date of disease progression (PD) or to death. Patients without PD who discontinued the study for any reason is censored at the last on-study tumor assessment date.
overall survival | 3 years
  OS and MST will be calculated from randomization to death from any cause or the date of the last follow-up, at which point the data will be censored.
tumor response | 3 years
  defined as partial and complete response according to RECIST 1.0 (Response Evaluation Criteria in Solid Tumors).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ye LC, Liu TS, Ren L, Wei Y, Zhu DX, Zai SY, Ye QH, Yu Y, Xu B, Qin XY, Xu J. Randomized controlled trial of cetuximab plus chemotherapy for patients with KRAS wild-type unresectable colorectal liver-limited metastases. J Clin Oncol. 2013 Jun 1;31(16):1931-8. doi: 10.1200/JCO.2012.44.8308. Epub 2013 Apr 8. PMID 23569301